CLINICAL TRIAL: NCT00315523
Title: Double-blind, 3 Parallel Randomized Groups, Therapeutic Confirmatory. Clinical Trial to Compare the Efficacy of Levocetirizine 5 mg and Montelukast 10 mg to Placebo in Reducing SAR Symptoms in Ragweed Sensitive Subjects in an EEC.
Brief Title: Compare the Efficacy of Levocetirizine to Montelukast in Reducing Symptoms of SAR in Sensitive Subjects Exposed to Ragweed Pollen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00415
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-05

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Levocetirizine; Xyzal; Rhinitis; Allergic; Seasonal; Ragweed
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — levocetirizine

INTERVENTIONS:
Drug: Levocetirizine

SUMMARY:
To compare the clinical efficacy of levocetirizine 5 mg and montelukast 10 mg, administered once daily during two consecutive days, on symptoms of seasonal allergic rhinitis occurring in subjects exposed to ragweed pollen in an environmental exposure unit.

ELIGIBILITY:
Inclusion Criteria:

* Have had seasonal allergic rhinitis due to Ragweed for the last 2 consecutive years
* Subjects who obtain a minimum sum score, considering SAR related symptoms (mean value), as defined by the protocol

Exclusion Criteria:

* Any clinically significant condition that might interfere with the treatment evaluation, both for efficacy and safety
* Have used forbidden concomitant medications as defined by the protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 403
Dates: Start 2006-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of Levocetirizine 5 mg to montelukast 10 mg as measured by the mean change from baseline of major symptoms related to SAR in ragweed sensitive subjects.

SECONDARY OUTCOMES:
Reduction in other SAR symptoms at different time points; Safety .

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Patel P, Patel D. Efficacy comparison of levocetirizine vs montelukast in ragweed sensitized patients. Ann Allergy Asthma Immunol. 2008 Sep;101(3):287-94. doi: 10.1016/S1081-1206(10)60494-2. PMID 18814452